## **INFORMED CONSENT FORM (ENGLISH)**

| Reg. No: | |
|---|---|
| I, Mr./Ms./Mrs | do hereby state willingly that I have been briefly |
| explained about the details of this clinical | ll research project entitled as "Synergistic effect of Vitamir |
| E and Vitamin D in reducing risk | of side effects associated typical anti psychotics and |
| improvement of psychiatric illness", | which is being undertaken by Dr.Mohammad Abid. I do |
| hereby give my written consent to get m | nyself registered in this study after considering the potentia |
| benefits that it will offer to the health | care services for the general public without any monetary |
| settlements. | |
| Participant's Signature: | |
| Date: | |
| Researcher's Signature: | |
| Date: | |

## **INFORMED CONSENT FORM (URDU)**

## راضى نامہ

اس تحقیقی کام میں شرکت کرنے کے لئے آپکا بہت شکریہ اگر آپ اس کام میں شامل ہورہے ہیں تو آپکو 5 ملی لیٹرخون کانمونہ دینے کو کہا جائیگا جو کہ ایک تجربہ کار ڈاکٹر سرنج کے ذریعے لیے گا۔ یہ نمونہ لیبارٹری میں محفوظ کیا جائے گا۔ خونکالنے سے کسی قسم کا کوئی نقصان نہیں ہوگا ۔ بعد ازاں یہ نمونہ تحقیق کے لئے استعمال کیا جائے گا۔ یہ تحقیقی کام کسی کاروباری مقصد کے لئے نہیں ہے۔ آپکی شمولیت آپکی مرضی پر ہے اور آپ کسی بھی وقت اس تحقیق سے الگ ہوسکتے ہیں آپ سے حاصل ہونے والی تمام معلومات کو صیغہ راز میں رکھاجائے گا اور یہ معلومات صرف تحقیق کرنے والوں کو میسر ہونگی۔ اگر اس تحقیق کے نتائج سے صحت کے متعلق نئی سائنسی معلومات حاصل ہوئیں تو وہ آپکے نام کو ظاہر کئے بغیر سائنسی جریدے یا رسالے میں شائع کی جائیگی۔ اس خون کے نمونے سے اس کے علاوہ کوئی کام نہیں لیا جائے گا۔

میں تصدیق کرتا /کرتی ہوں کہ میں نے اس دستاویز کو سمجھ لیا ہے میں اپنی مرضی سے اپنے میں اپنی مرضی سے اپنے خون کا نمونہ اس تحقیقی کام میں دینے کے لئے تیار ہوں۔

| ستخط: | نام مریض: ۔۔۔۔۔۔۔۔۔۔ د |
|--------|-----------------------------|
| تاريخ: | راضى نامم لينسر والسركا نام |